CLINICAL TRIAL: NCT06293716
Title: An Open, Dose-exploration Study, Followed by a Randomized, Double-blind, Placebo-controlled Study, to Evaluate the Efficacy and Safety of CVL237 Tablets in Patients With APDS/PASLI
Brief Title: CVL237 Tablets for APDS/PASLI
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Convalife (Shanghai) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CVL237-A2001
Record Dates: First submitted 2024-02-18; First posted 2024-03-05 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-02

CONDITIONS: PI3K and P110delta Hyperactivation Syndrome
Keywords: PI3K; P110delta; hyperactivation
MeSH Terms: conditions — Hereditary Sensory and Autonomic Neuropathies

STUDY DESIGN:
Intervention Model Description: CVL237 tablets for APDS/PASLI (Activated phosphoinositol 3-kinase delta syndrome /p110 delta-activated Mutation leading to senescent T cells, lymphadenopathy, and immune deficiency)
Who Masked: Participant, Investigator
Masking Description: Part II is a randomized, double-blind, placebo-controlled study of approximately 30 patients with APDS/PASLI. On day 1, patients were randomly assigned to the trial and placebo groups in a 2:1 ratio to take an oral CVL237 tablet or a placebo CVL237 simulant once daily. Efficacy and safety were evaluated on days 29, 57, and 85. The efficacy of CVL237 tablets in reducing lymphadyopathy will be investigated as measured by changes in the sum of diameter products (SPD) of target lesions selected from MRI or CT imaging according to the Lugano 2014 method, as well as changes in the percentage of naive B cells to total B cells, relative to baseline. The CVL237 tablets will also be evaluated for safety, PK
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- part1:treatment group (Experimental): Patients were given CVL237 tablets, 100 mg/ day, QD, for 4 weeks (28 days), and safety assessment was performed on day 28 of the first cycle. If there was no safety risk, patients could take CVL237 tablets, 200 mg/ day, QD, for 4 weeks (28 days).
  Interventions: Drug: CVL237 tablets
- part2:treatment group (Experimental): Patients were randomly assigned to the trial and placebo groups in a ratio of 2:1 to take an oral CVL237 tablet once daily.
  Interventions: Drug: CVL237 tablets
- part 2:placebo group (Placebo Comparator): Patients were randomly assigned to the trial and placebo groups in a ratio of 2:1 to take a placebo CVL237 simulant once daily.
  Interventions: Drug: CVL237 placebo tablets

INTERVENTIONS:
Drug: CVL237 tablets — CVL237 tablets, tablets, specification: 0.1g, Storage condition: not more than 30 ℃ storage.Validity: 72 months tentatively.
  Arms: part1:treatment group; part2:treatment group
Drug: CVL237 placebo tablets — CVL237 tablets, tablets, specification: 0g, Storage condition: not more than 30 ℃ storage.Validity: 72 months tentatively.
  Arms: part 2:placebo group

SUMMARY:
This study was designed to evaluate the efficacy and safety of CVL237 tablets in patients with APDS/PASLI (activated phosphoinositol 3-kinase δ syndrome /p110 delta-activated mutation leading to senescent T cells, lymphadenopathy, and immune deficiency).

DETAILED DESCRIPTION:
The study was divided into two parts.

Part I is an open, dose-escalation study planned to enroll five patients with APDS/PASLI to determine the safety, tolerability, pharmacokinetics (PK), and in vivo pharmacodynamics (PD pAkt) of CVL237 tablets at two different dose levels. Patients were given CVL237 tablets, 100 mg/ day, QD, for 4 weeks (28 days), and safety assessment was performed on day 28 of the first cycle. If there was no safety risk, patients could take CVL237 tablets, 200 mg/ day, QD, for 4 weeks (28 days).

Part II is a randomized, double-blind, placebo-controlled study of approximately 30 patients with APDS/PASLI. On day 1, patients were randomly assigned to the trial and placebo groups in a 2:1 ratio to take an oral CVL237 tablet or a placebo CVL237 simulant once daily. Efficacy and safety were evaluated on days 29, 57, and 85. The efficacy of CVL237 tablets in reducing lymphadyopathy will be investigated as measured by changes in the sum of diameter products (SPD) of target lesions selected from MRI or CT imaging according to the Lugano 2014 method, as well as changes in the percentage of naive B cells to total B cells, relative to baseline. The CVL237 tablets will also be evaluated for safety, PK.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients aged 18-75 years (including boundary values);
* Patients with a clinical phenotype consistent with APDS, including a history of recurrent ear, sinus, or lung infections (more frequently than expected in immunoactive individuals), and patients known to have type 1 APDS-related gene PI3K mutations (e.g., E1021K, N334K, E525K, and C416R) or type 2 APDS-related mutations;
* In Parts I and II, the patient must have lymph node and/or extranodal lymphocyte proliferation, as well as clinical findings and manifestations consistent with APDS/PASLI, such as a history of recurrent ear - sinus - lung infections and/or organ dysfunction (e.g., lung, liver). In addition, in Part II, patients must have at least one measurable lymph node lesion on a CT or MRI scan.
* During screening, vital signs (systolic blood pressure, diastolic blood pressure, and pulse rate) were assessed by sitting position after at least 3 minutes of rest. Seated vital signs should be within the following range:
* Systolic blood pressure, 90-139 mm Hg
* Diastolic blood pressure, 50-89 mm Hg
* pulse rate, 50-100 bpm; Up to 110 bpm in teenagers
* Expected survival ≥3 months;
* Pregnant or lactating women or fertile women with a negative pregnancy test at baseline; Men and women with 6) fertility must consent to the use of medically approved contraceptive methods during the study period and within 6 months after the last dosing;
* Did not participate in any clinical trials within 1 month before joining the study;
* Able to comply with the test protocol (as determined by the investigator);
* Volunteer to participate in this clinical trial, understand the study procedure and be able to sign the informed consent in person.

Exclusion Criteria:

* Previous or concurrent use of immunosuppressive drugs, such as:

  1. Use of mTOR inhibitors (e.g., sirolimus, rapamycin, Everolimus) or PI3kδ inhibitors (selective or non-selective PI3K inhibitors) within 5 half-lives prior to initial medication, but allow short-term use, for a total of no more than 5 days, but only within 1 month prior to enrollment in the study.
  2. Use B cell depleting agents (e.g. Rituximab) within 5 half-lives prior to initial administration; If the patient has previously been treated with B cell depleting agents, the absolute B lymphocyte count in the blood must return to normal.
  3. had taken Belimumab or cyclophosphamide within 5 half-lives before first taking the study drug.
  4. Use of cyclosporin A, nystatin, 6-mercaptopurine, azathioprine, or methotrexate within 5 half-lives prior to first administration of the study drug.
  5. Use more than 25 mg of prednisone or an equivalent dose of glucocorticoids daily for 2 weeks prior to the first dose.
  6. Other immunosuppressive drugs whose effects are expected to remain at the start of the study.
* Being treated with known OATP1B1 and OATP1B3 substrate drugs, CYP3A4/5 substrate drugs, intermediate-acting and potent CYP3A4/5 inhibitors, CYP3A4/5 potent inducers, if treatment cannot be terminated or switched to another drug before initiating investigational therapy;
* Drugs currently used that are metabolized by the isoenzyme CYP1A2 and have a narrow therapeutic index (exposure responses indicate that drugs that accompany increasing their exposure levels with the use of powerful inhibitors may cause serious safety concerns (e.g., tip torsion ventricular tachycardia))
* Current history of liver disease or chronic disease, unless liver enlargement is determined by their clinicianto be secondary to APDS, or known liver or biliary tract abnormalities (other than Gilbert syndrome or asymptomatic gallstones)
* The investigator determined that the patient had clinically significant abnormalities in laboratory results (blood routine, blood biochemical, or urine routine)
* Patients with liver disease or liver injury, clinically significant abnormal liver function tests (alanine aminotransferase and aspartate aminotransferase > 2.5 times the upper limit of normal), a history of kidney injury/kidney disease (e.g., kidney trauma, glomerulonephritis, or having only one kidney), or impaired kidney function, The serum creatinine level was >1.5 mg/dL (133 μmol/L). LVEF < 50%, Fridericia corrected QT Interval (QTcF) ≥450 ms for men and 470 ms for women;
* If a subject's clinical abnormality or laboratory parameters are not specifically listed in the inclusion or exclusion criteria and are outside the reference range of the studied population, they may be included in the study only if the investigator agrees and records that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedure.
* The history of regular alcohol consumption within 6 months of the study was defined as an average weekly intake of > 14 units. One unit is equivalent to 8 grams of alcohol: half a pint (~240 ml) of beer, 1 glass (125 ml) of wine or 1 glass (25 ml) of spirits.
* Screen positive for substance abuse. Testing for drugs used for legitimate medical purposes (e.g. benzodiazepines, opioid analgesics) does not necessarily exclude study participation and will be at the discretion of the principal investigator.
* A history of sensitivity to any investigational drug or its components (including lactose) or to a history of drug or other allergies (including milk protein allergies) that the investigator deemed unsuitable for participation in the study.
* Positive hepatitis B surface antigen (HBsAg) and hepatitis C antibody test results at the time of screening or within 3 months before first receiving the study drug. Patients infected with hepatitis B virus (HBV) or hepatitis C virus (HCV) (defined as Hepatitis B Surface antigen (HbsAg) and/or Hepatitis B core antibody (HbcAb) positive and HBV DNA > 500 IU/mL or > 2500 copies/mL; Positive anti-HCV antibody and HCV-RNA quantification > upper limit of normal test unit).
* Have uncontrolled pulmonary fibrosis, acute lung disease, interstitial pulmonary inflammation;
* People with active viral, bacterial, fungal or other infections requiring systematic treatment (e.g., active tuberculosis), excluding nail bed fungal infections;
* Blood donation/blood loss ≥400 ml or more within 8 weeks before the first dose;
* History of immunodeficiency (acquired and congenital), history of organ transplantation, allogeneic bone marrow or hematopoietic stem cell transplantation; Active autoimmune disease or history of autoimmune disease (such as autoimmune enteritis and systemic lupus erythematosus);
* There are many factors affecting drug administration and absorption, such as inability to swallow, chronic diarrhea, intestinal obstruction (functional).
* Participants participated in a clinical trial and received the investigational drug during the following time period prior to administration of the first investigational drug in this study: 30 days, 5 half-lives, or twice the duration of the investigational drug's biological effect, whichever is older.
* Present with difficult or important cardiovascular disease: history of heart or aortic surgery; History of myocardial infarction; Had uncontrollable angina in the 6 months prior to the screening period, or is currently taking anti-angina medication; Grade III/IV congestive heart failure; Arrhythmias requiring clinical intervention; Any other cardiovascular disease that the investigator determines is not suitable for participation in the study;
* Live vaccines (including any attenuated live vaccines) were administered within 6 weeks before the first administration of the trial drug, during the study period and within 7 days after the last administration of CVL237 tablets.
* Patients who cannot stop taking medications that may cause QT prolongation, such as antiarrhythmic drugs, during the study period.
* The patient has a history of malignancy (other than lymphoma) or evidence of residual disease from a previously diagnosed malignancy within 3 years prior to initial dosing;
* Subjects deemed unsuitable for this trial for other reasons.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2024-03-30 (Estimated); Primary Completion 2025-12-29 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
part 1 : Incidence of Treatment-Emergent Adverse Events | Throughout the study for approximately 84 days
  Abnormal changes in physical examination, vital signs, electrocardiograph laboratory tests, etc. compared to baseline were reported as AE
part 2:After 84 days of treatment, changes in the sum of diameter product (SPD) of log10 conversion in target lesions and changes in the percentage of naive B cells to total B cells from baseline were observed | At baseline (day 0) and at the end of treatment (day 84)
  SPD:The maximum diameter of the tumor is multiplied by the longest diameter perpendicular to it

SECONDARY OUTCOMES:
Cmax | part 1： Up to day 56；part 2： Up to day 85
  Peak concentration: The highest blood concentration after administration
t1/2 | part 1： Up to day 56；part 2： Up to day 85
  Terminal elimination half-life: The time required for the terminal phase blood concentration to decrease by half
AUC | part 1： Up to day 56；part 2： Up to day 85
  Area under the drug time curve: The area surrounded by the blood concentration curve to the time axis.
Tmax | part 1： Up to day 56；part 2： Up to day 85
  Peak time: The time required to reach peak concentration after administration

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Public Health Clinical Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No